CLINICAL TRIAL: NCT02226029
Title: Quantitative Magnetic Resonance (MR) Methods for Non-invasive Imaging of Gastro-intestinal (GI) Processing of Lipid Emulsions in Healthy Subjects.
Brief Title: Quantitative MR Methods for Lipid Emulsions
Acronym: Q-MRemulsion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: KEK-ZH-Nr. 2014-0185; SNF #146409 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: MRI, fat fraction, stomach, lipid emulsion
MeSH Terms: interventions — Fat Emulsions, Intravenous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lipid emulsion 1 (Experimental): Rapeseed oil 20%, sucrose FAE P-1670 0.7%, water 79.3%
  Interventions: Other: Lipid emulsion
- Lipid emulsion 2 (Experimental): Rapeseed oil 20%, sodium stearoyl lactylate P45 veg 1.5%, water 78.5%
  Interventions: Other: Lipid emulsion

INTERVENTIONS:
Other: Lipid emulsion — 2 isovolumetric (200 ml) and isocaloric (200 kcal) lipid emulsions with different acid and shear stability
  * Lipid emulsion 1: acid stable, particle size 0.6 µm
  * Lipid emulsion 2: acid unstable, redispersible by mechanical processes during antral contractions and passage through the pylorus, particle size 0.6 µm
  * 13C-markers will be mixed with emulsions

SUMMARY:
Quantitative MR methods will be validated for the non-invasive imaging of GI processing of lipid emulsions in 18 (12+6) healthy subjects. Validation is performed by a randomized single blind two-armed crossover trial with two isovolumetric and isocaloric lipid emulsions of different microstructural properties. Hypotheses of this sudy are that

1. the fat fraction of lipid emulsions in the GI tract can be monitored by quantitative MR methods and that 13C-sodium octanoate and
2. 13C-sodium acetate in lipid emulsions will exhibit different excretion profiles due to their opposing binding affinity to water and fat.

DETAILED DESCRIPTION:
Participants will be given two lipid emulsions with different physicochemical composition in randomized order at two separate visits. A nasogastric tube will be applied for intragastric lipid emulsion infusion to control for the effect of inter-individual tolerance to texture and taste of the lipid emulsions. Standard MR measurements will be performed to regularly assess intragastric fat content and related fat content emptying over a period of 3 hours. At different pre-defined time points during gastric processing and emptying of the emulsions, five samples of gastric content (5x2 ml) will be aspirated via the nasogastric tube to determine local intragastric fat content with a density measurement. The measured fat fraction of the aspirated samples will validate the non-invasive quantitative MR measurements. Each participant will also undergo either a 13C-sodium acetate or a 13C-sodium octanoate breath test at each of the two visits. Breath tests will be carried out throughout the MR imagining period and for 2 hour post imaging. A subset of participants will undergo the same breath test procedures but without the use of MR and gastric content samples.

2 isovolumetric (200 ml) and isocaloric (200 kcal) lipid emulsions with different acid and shear stability. 13C-markers will be mixed with emulsions.

* Lipid emulsion 1: acid stable, particle size 0.6 µm
* Lipid emulsion 2: acid unstable, redispersible by mechanical processes during antral contractions and passage through the pylorus, particle size 0.6 µm

Power calculation is based on an in-vitro pilot experiment, in which we determined a variation in the detection of fat fraction in the lipid emulsions of 1.5%. With 12 enrolled subjects, the detectable difference in fat fraction at a significance level of 0.05 and a defined power of 0.9 is about 2%. In 18 enrolled subjects (12+6) that are separated into two groups of 9, the detectable difference in 13CO2 recovery at a significance level of 0.05 and a defined power of 0.9 is 0.15 Percent Dose Recovered per hr (PDR/hr).

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP or ISO EN 14155 (as far as applicable) as well as all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between age 18 and 50
* BMI 18-25 kg/m²
* Written informed consent

Exclusion Criteria:

* History of GI, cardiorespiratory (including arterial hypertension), hematologic, renal, atopic, alimentary or psychiatric disorder, panic attacks, diabetes, drug or alcohol abuse
* Prior abdominal surgery other than uncomplicated appendectomy or hernia repair
* Requiring medication that might alter gut function, including anticholinergics, calcium channel blockers, beta blockers, laxatives, prokinetics, proton-pump inhibitors, non-steroidal anti-inflammatory drugs
* Presence of metallic implants, devices or metallic foreign bodies
* Pregnancy and lactation (female participants of child bearing age will receive a pregnancy test prior to study)
* Claustrophobia
* Regular smoking or consumption of alcohol and drugs
* Uncertainty about the willingness or ability of the participant to comply with the protocol requirements

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Fat fraction [%] of GI content | up to 180 minutes

SECONDARY OUTCOMES:
Distal fat fraction [%] | 3, 10, 20, 30, 45, 60, 90, 120, 150 and 180 minutes

OTHER OUTCOMES:
Parameters k and β from model B(t) = Dose*[β*(1- e(-k *t))(β-1) - (β- 1)*(1- e(-k *t))β] fitted to the 13C excretion profiles | every 10 minutes until 300 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Steingötter, PhD, Principal Investigator — University of Zurich
Locations (1):
- Division of Gastroenterology and Hepatology, University Hopsital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Parker HL, Liu D, Curcic J, Ebert MO, Schwizer W, Fried M, Steingoetter A. Gastric and Postgastric Processing of 13C Markers Renders the 13C Breath Test an Inappropriate Measurement Method for the Gastric Emptying of Lipid Emulsions in Healthy Adults. J Nutr. 2017 Jul;147(7):1258-1266. doi: 10.3945/jn.117.248765. Epub 2017 May 31. PMID 28566523